CLINICAL TRIAL: NCT03557528
Title: Evaluation of the Role of Low Inferior Mesenteric Artery Ligation During Laparoscopic Surgery for Rectosigmoid Tumors
Brief Title: Role of Low Inferior Mesenteric Artery Ligation During Laparoscopic Surgery for Rectosigmoid Cancer
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, DANIELE CROCETTI, MD, PhD, University of Roma La Sapienza
Other Study IDs: 14ur2018
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Rectosigmoid Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: High Ligation of Inferior mesenteric artery
  Interventions: Procedure: Laparoscopic colorectal resection
- Group 2: Low ligation of inferior mesenteric artery with skeletonization at its origin
  Interventions: Procedure: Laparoscopic colorectal resection

INTERVENTIONS:
Procedure: Laparoscopic colorectal resection — Gruop 1: laparoscopic rectosigmoid resection with standard ligation of mesenteric artery at its origin Group 2: Laparoscopic rectosigmoid resection with low ligation of inferior mesenteric artery and its skeletonization with en bloc removal of all lymph nodes

SUMMARY:
During sigmoid or rectal cancer surgery, dissection of lymphnodes at the origin of inferior mesenteric artery is mandatory. Nevertheless, ligation of the origin of IMA should compromise blood supply to left colon and affect anastomosis. The aim of this retrospective evaluation is to compare high and low IMA ligation with preservation of LCA, with or without skeletonization of the origin of IMA in laparoscopic colorectal resection.

ELIGIBILITY:
Inclusion Criteria:

* stage I-III carcinoma

Exclusion Criteria:

* stage IV
* Urgent resection
* conversion to open surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients affectced by clinical stage I-III cancer of sigmoid and rectum.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
effectivenes of lymphnode dissection | 3 years
  number of dissected lymphnodes

SECONDARY OUTCOMES:
complication | 3 years
  incidence of anasthomotic leaks

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I, Roma, Italy

IPD SHARING:
Plan to Share IPD: No